CLINICAL TRIAL: NCT01411605
Title: Influence of Cardio-ventilatory Factors on Exercise Intolerance in Obese Adolescents: Effects of Exercise Training
Acronym: VENTILOBE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0718; 2007-A00714-49 (Registry Identifier: ID RCB)
Record Dates: First submitted 2011-07-29; First posted 2011-08-08 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Obesity
Keywords: Obesity; Adolescent; Exercise training; Exercise tolerance
MeSH Terms: conditions — Obesity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise training (Experimental): 12-week supervised exercise-training (ET) program consisting of two 60-min and one 120-min exercise sessions per week which focus mainly on aerobic exercises (cycling, treadmill, rower).
  Initial aerobic exercise intensity is set at 60 % of HR peak and will reach 80 % at the end of the ET protocol.
  Interventions: Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Exercise training — 12-week supervised exercise-training (ET) program consisting of two 60-min and one 120-min exercise sessions per week which focus mainly on aerobic exercises (cycling, treadmill, rower).
  Initial aerobic exercise intensity is set at 60 % of HR peak and will reach 80 % at the end of the ET protocol.

SUMMARY:
Worldwide, childhood and adolescent obesity has reached epidemic proportions despite major efforts to promote weight reduction. Pediatric obesity commonly presages adult obesity and is associated with the development of weight-related comorbid conditions and increased morbidity.

Regular physical activity is an important modality of obesity management. Despite controversies, poor exercise tolerance has frequently been reported in youth obesity and the cause of this limited exercise tolerance remains unknown. Several factors accompanying obesity may interfere with exercise tolerance in obese populations. Respiratory factors, such as decreased thoracic compliance, increased airway resistance and breathing at low pulmonary volumes are associated with obesity and may impact exercise intolerance in this population. Moreover, even in people with otherwise normal lungs, the normal ventilatory responses to exercise can become constrained in obesity. A thorough understanding of the mechanisms underlying this exercise intolerance remains fundamental in order to favour long term adherence to exercise training. This is especially true in youth populations, in which the management of overweight and obesity must be undertaken as soon as possible, due to the early onset of cardiovascular risk factors.

The main purpose of this study is to determine early-onset cardio-respiratory mortality factors in obese adolescents as well as their relation with exercise intolerance (i.e. dyspnea) when compared with age and gender-paired normal-weight volunteers.

DETAILED DESCRIPTION:
Physiopathological trial. Expected total enrollment : 20 obese adolescents + 20 control subjects Tested treatment: Exercise training (4 hours per week). Treatment duration: 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* Male and female obese adolescents (BMI > IOTF 30, 12-16 years old)

Exclusion Criteria:

* Cardiovascular pathology
* Pathology interfering with physical activity (neurological pathology, severe respiratory illness i.e. asthma, renal failure)
* Diabetes (known or treated)
* Participation in another study
* Asthma (known and treated)

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2007-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Exercise tolerance (Expiratory flow limitation and Operational Lung Volumes at rest and exercise, cardiorespiratory and subjective responses to incremental exercise) | Participants will be followed for the duration of exercise training, an expected average of 12 weeks

SECONDARY OUTCOMES:
Polysomnography | Participants will be followed for the duration of exercise training, an expected average of 12 weeks
  Explore the potential existence of obstructive sleep apnea and its effects on cardiovascular adaptations during exercise.
Cardiorespiratory fitness (VO2max) | Participants will be followed for the duration of exercise training, an expected average of 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bernard WUYAM, Dr, Principal Investigator — University Hospital, Grenoble; Claudine Perrin, MD, Principal Investigator — CHU Grenoble, Pediatrics Department
Locations (1):
- CHU Grenoble, Grenoble, France